CLINICAL TRIAL: NCT06616935
Title: Routine Referrals to Third Sector Organisations Following Reablement to Target Loneliness Among Older Adults Aged 65years and Over.
Brief Title: Beyond Older Adults' Reablement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Northampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DCaesar Reablement
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2024-09

CONDITIONS: Loneliness
Keywords: Loneliness; Older Adults; Reablement; Intermediate Care

STUDY DESIGN:
Intervention Model Description: Intervention one: community activities. Intervention two: online exercises and activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine referrals to community activities (Other): Routine referrals to community activities following receiving reablement and being discharged without further action.
  Intervention group 1 referrals to community activities.
  Interventions: Other: Intervention group one, community activities.
- Online exercises and activity (Other): Online exercises and activity group.
  Interventions: Other: Intervention group two

INTERVENTIONS:
Other: Intervention group one, community activities. — Intervention group one: participants will have a list of free activities in the community provided by third sector organisations to choose from. Participants will be referred to their chosen activities and expected to attend for six months.
  Intervention group two: Participants will attend weekly online exercises and activities led by the researcher.
  Arms: Routine referrals to community activities
Other: Intervention group two — Online exercises and activities
  Arms: Online exercises and activity

SUMMARY:
The goal of this feasibility study is to find out if routine referrals of older adults aged 65years and over to community activities provided by third sector organisations will reduce their loneliness risk.

Researcher will compare referrals of older adults to community activities following reablement provided by intermediate care to attendance of online activities to find out which will be effective in reducing loneliness risk of older adults aged 65years and over. Researcher will also find out if it will be feasible to complete a full randomised controlled trial.

DETAILED DESCRIPTION:
Introduction The older adult population is increasing in England and Wales. In 2001, there were 8.3million aged 65years and over compared to 11million in 2021. This has resulted in their increased hospital admissions with subsequent use of reablement following discharge. Older adults will be used to represent those aged 65years and over for this study.

Reablement aims at increasing independence of older adults and is being used to reduce their care cost. However, there is an apparent contradiction in that many older adults are often socially isolated following an episode of reablement. Loneliness has also been reported among older adults and this has the potential of impacting on their psychological and physical wellbeing.

This research will investigate the impact of routinely referring older adult reablement recipients to services in the community (neither public nor private sector) known as third sector organisations (National Audit Office) that target loneliness to reduce their recurrent admissions to hospitals. It will be carried out in an Intermediate Care Team providing reablement in the East Midlands of England. Background Reablement is a short-term (up to six weeks) programme aimed at relearning skills that are lost through ill health. Locally, Intermediate Care Team (ICT) of the National Health Service (NHS) facilitates and prevents admissions from hospitals by providing reablement at the home of patients in the County being studied. ICT is however, commissioned to discharge patients within 17 days of admission to its caseload. It is not clear whether reablement programmes are set to address longer-term issues of recipients during and after the service. Support systems after the service of those who emerge independent are also not clear. These were noted from a service evaluation carried out by the researcher and other researchers have also note the paradoxical increase in hospital admissions following reablement of older adults. These could be related to the psychological and physical factors affecting recipients who emerge independent and end up living alone with no services involved. Literature Review There is a plethora of literature on the positive impacts of reablement on the physical abilities of older adults. Older adult recipients find it beneficial, and report increase independence of their activities of daily living . Some recipients have also been reported to have reduced home care leading to reduction in financial cost of care. Positive mental wellbeing and social functioning of some recipients have been reported.

There is, however, a paucity of literature on the impact of loneliness on older adults who receive reablement, particularly those who are discharged as independent but have no family support. As reablement promotes independent living, there could be a possibility of some recipients being at risk of loneliness and isolation. efficient ways of maintaining the quality of life of older adults is needed amidst the increase in the older adult population and budget cuts of local governments. In studies to find out the effectiveness of interventions to reduce loneliness among older adults, their active participation in group activities has been found to limit their loneliness. Other studies however, did not find group interventions more effective compared to one- to- one interventions in tackling older adults' loneliness. Some studies also did not find social intervention effective in reducing loneliness. Video conferencing has been found effective in directly and indirectly reducing loneliness among older adults but has its own limitations of health inequalities.

Social prescribing helps patients access nonclinical support . This is however mainly available through some General Practitioner (GP) services. The older adult patients described in this study might likely not be accessing such support. The Innovation Potential This study will ascertain third sector organisations currently available in the community for older adults deemed as independent after receiving reablement with stakeholders. It will explore whether these services are sufficient or appropriate to meet the needs of older adults who are socially isolated and at risk of loneliness. Older adults will be involved in the development of the project to identify solutions. This will add to the evidence base for longer-term impact beyond the initial reablement episode. Aim To find out whether routine referrals to third sector organisations of older adults who have been discharged as independent from ICT will be effective in reducing their loneliness risk and recurrent hospital admissions. Objectives Objective 1: To complete a literature review on older adults' loneliness and reablement. Objective 2: To identify third sector organisations available in the local area for socially isolated older adults. Objective 3: To co design questions for semi structured interviews of older adult ICT patients to be referred to the identified third sector organisations following reablement with an older adult Patient and Public Interest (PPI) group.

Objective 4: To conduct a feasibility study of routinely referring older adults to the identified third sector organisations with pre and post semi structured interviews following discharge from ICT to determine its effectiveness in reducing loneliness risk and recurrent hospital admissions. Objective 5: To estimate the rate of eligible older adults who are willing to participate, those who will drop out and those who will comply with the allocated intervention to assist in the design of a full randomised controlled trial. Research Design and Methods. This will be an applied health research employing empirical method. It will be mixed methods research of both quantitative (feasibility) and qualitative (semi structured interviews) methods in five phases. The phases will be literature review, service mapping, followed by a participatory action research (PAR) approach to co design questions for the semi structured interviews for participants in the feasibility study phase. The feasibility study will be to implement outcomes from the second and third phases for effectiveness and feasibility for a larger scale randomised controlled trial. A sample of the participants will be interviewed pre and post the interventions for triangulation (Hussein, 2009). The final phase will be estimation of the rate of eligible participants willing to participate, those who will drop out and those who will comply with the intervention to assist in designing a full randomised controlled trial. A pragmatism epistemology will be assumed to allow a co-produced solution to the research question. Setting Reablement service provided through ICT in the East Midlands of England due to the service facilitating discharges from hospitals but also experiencing recurrent admissions to its caseload. Process Phase one: Literature review A systematic approach of searching the literature through appropriate databases will be used to complete the literature review.

The literature will be reviewed on the definition of loneliness and its appropriate measurement with respect to older adults. The impact of loneliness on older adults and the interventions for tackling loneliness among older adults will also be reviewed. Reablement being provided in facilitating and preventing hospital admissions will also be reviewed. Phase two: Service mapping exercise. The public health departments of the county being studied will be contacted to get information on the available services for older adults in the community. The local Age United Kingdom (UK), charity services, Church of England churches, Salvation Army churches, Baptist churches, libraries, Caribbean Groups, African groups, Asian Groups, Sikh Community will also be contacted for information on their available services. These have been identified as stakeholders in older adult care in the county. Therapy colleagues from the workplace will also be engaged for their input on available services within the county.

Phase three:

Co Designing with Patient and Public Interest (PPI) Group A Participatory Action Research (PAR) approach has been employed to engage a PPI group. The PPI group was made of four older adults and were consulted on a one-to-one basis. The PPI group helped in developing the questions to be asked in the semi structured interviews. This is to allow a co-production of the questions for the semi structured interviews for the feasibility phase. The Research Development Service (RDS) advocates the involvement of PPI group in health research as they would have a better experience of what is being researched. Studies have shown that older adults wish to be involved in project development and delivery. Interventions that involve users in design and implementation are more successful.

Phase four:

Feasibility Study (Quantitative study) Older adults about to be discharged from ICT independently, faced with loneliness will be approached for participation. Potential participants who show interest and give informed written consent will have the 11 item De Jong Gierveld loneliness scale administered to identify their loneliness risk. This has been chosen over the 3 item University of California Los Angeles (UCLA) loneliness scale as it measures items specific to the research with respect to isolation and loneliness. Those identified as at risk of loneliness (score of at least 3) will be included in the study and those not at risk will no longer be included. They will then be assigned randomly to the intervention groups using sealedenvelope.com. The researcher who is also the chief investigator will have no access to the allocation sequence.

Participants in the intervention one group will have a choice of the activities in the community they would like to attend. Participants in the intervention two group will attend weekly online seated and standing exercises and discussions via TEAMS led by the researcher. Participants' physical and mental wellbeing will be measured with the EQ-5D-5L scale and demographic data of age, sex, ethnicity, marital status and whether they have family will be taken. Their frailty Index score will be noted pre and post the study. These will help gain background information about the participants.

Semi Structured Interviews (Qualitative Study) Semi structured interviews will be conducted with some randomly selected participants from both groups pre and post intervention. The interviews are expected to last for up to one hour and will be recorded with a password protected audio recorder.

Phase five:

Estimating the participating rate. The number of participants willing to take part, those who will drop out, comply with the interventions, and sample size for the actual randomised controlled trial will be determined.

Data analysis The interviews will be organised using NVivo 12 and analysed using thematic analysis to obtain the main themes. Two-way ANOVA (Analysis of Variance), intervention one group verses intervention two group and pre-test verses post-test will be conducted using SPSS software to analyse data from the feasibility study. Demographic data will also be analysed with the SPSS software. The participating rate, sample size as well as the standard deviation of the main outcome measure De Jong Gierveld Loneliness scale will be determined for the actual randomised controlled trial. Hypothesis to be tested.

1. There is no difference in the De Jong Gierveld loneliness scores between older adults who attended community activities for six months and those who attended online activities for six months.
2. There is no difference in EQ 5L 5D scores between older adults who attended community activities for six months and those who attended online activities for six months.
3. There is no difference in the frailty scores between older adults who attended community activities for six months and those who attended online activities for six months.

Ethical Considerations Permission to complete the study will be sought from ICT managers. Ethical approval will be sought from the Integrated Research Application System (IRAS), Health Research Authority (HRA), and the University of Northampton Ethics Committee.

Potential Participants will be issued Participant Information Sheets and given seven days to read, understand and ask questions. The participant information sheet has been checked by two older adults for language and clarity.

Informed written consent will be sought from participants prior to taking part in the study and they will be informed of their right to withdraw up to the data analysis stage through the participant information sheets without repercussions according to the declaration of Helsinki (World Medical Association, 2013). Participants who will be selected for the semi structured interviews will have to sign a second consent form specific to the interview.

Participants' data will be anonymised to remove identifiable information for their confidentiality. The data will be stored securely in accordance with the General Data Protection Regulation (GDPR) 2018 in the University of Northampton's SharePoint.

ELIGIBILITY:
Inclusion Criteria:

* Past and current patients of the team aged 65years and over retrieved from 12months up to the month of recruitment (August 2023 to September 2024).
* Patients who have had at least three hospital admissions and three admissions to the team.
* Patients whose admissions resulted or will result in being discharged with no further action.
* Patients identified as at loneliness risk by a score of 3 or more on the De Jon Loneliness Scale.

Exclusion Criteria:

* Patients of the team who will be discharged with planned care package or family support.
* Patients of the team who lack mental capacity.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Risk of loneliness of participants as identified with the De Jon Gierveld (DJG)loneliness scale. | Enrollment where the initial measures will be taken and then at six months from when the initial measures were taken which will be the end of the study.
  Quantitative measure of loneliness risk from 0 (no risk) to 11(highest risk) with the DJG scale with a score of at least 3 representing being at risk of loneliness for the current study.
Frailty of participants as measured by the Frailty Index Scale. | Initial Frailty Index scale will be measured when participants are randomised to intervention groups and the final Frailty Index Scale will be measured six months from being assigned to intervention group.
  The Frailty Index Scale quantifies function between 1 and 9 with one being the least frail and 9 being very frail.
  This will help establish whether the intervention improves function in participants.
Self reported physical activity levels and mental wellbeing of participants as identified by EQ-5D-5L scale. | EQ-5D-5L will initially be collected when participants are randomised to intervention groups and again at six months from when they were randomised to intervention groups.
  The EQ-5D-5L scale is a self reported outcome measure which allows participants to assess their own physical function, mental wellbeing and health.
  This will help establish whether the interventions improve the reported physical function, mental wellbeing and health of participants or not.

SECONDARY OUTCOMES:
Feasibility Outcomes | Six months from enrolment where the outcome measures will be initially collected.
  1. Suitability of randomising participants.
  2. Feasibility of delivering the interventions within the time scale stipulated.
  3. Suitability and sensitivity of outcome measures to be used in a large trial.
Suitability of randomising participants as measured by the percentage of participants who will be able to attend their assigned interventions for the six month duration | The feasibility of randomising participants will be determined at six months from when participants were randomised to intervention groups.
  The suitability of randomising participants will help in planning an actual Randomized Controlled Trial in determining whether it will be appropriate to randomise participants to interventions. If only 10% of participants will adhere to their intervention group, it may not be suitable to randomise participants.
Feasibility of delivering the interventions within the time stipulated as identified by the percentage of participants completing their assigned interventions at six months from initial randomisation of participants. | The feasibility of delivering the interventions within the time stipulated will be determined at six months from the time of initial randomisation of participants to intervention groups.
  The feasibility of delivering the interventions will help in planning the actual time duration required in an actual Randomised Controlled Trial. If only 10% of participants are able to start and finish their assigned interventions from randomisation to the end of the interventions at six months, then the duration of the study may have to be extended.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Parkes, Professor, Study Director — University of Northampton Faculty of Health, Education &amp;amp;amp; Society
Locations (1):
- Intermediate Care Team, Kettering, Northamptonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This will be considered later.

REFERENCES:
- [Background] Gierveld, J. D. J., & Tilburg, T. V. (2006). A 6-item scale for overall, emotional, and social loneliness: Confirmatory tests on survey data. Research on aging, 28(5), 582-598.
- [Background] Findlay, R. A. (2003). Interventions to reduce social isolation amongst older people: where is the evidence? Ageing & Society, 23(5), 647-658.
- [Background] Clegg A, Bates C, Young J, Ryan R, Nichols L, Ann Teale E, Mohammed MA, Parry J, Marshall T. Development and validation of an electronic frailty index using routine primary care electronic health record data. Age Ageing. 2016 May;45(3):353-60. doi: 10.1093/ageing/afw039. Epub 2016 Mar 3. PMID 26944937
- [Background] Bartlett H., Warburton J., Lui C.-W., Peach L. & Carroll M. (2013). Preventing social isolation in later life: findings and insights from a pilot Queensland intervention study. Ageing & Society 33 (7), 1167-1189.
- [Background] Bowling, A., (2014). Research methods in health: investigating health and health services. McGraw-hill education (UK).
- [Background] Braun, V. Clarke, V. (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3 (2). pp. 77-101. ISSN 1478-0887 Available from: http://eprints.uwe.ac.uk/11735
- [Background] Aspinal F, Glasby J, Rostgaard T, Tuntland H, Westendorp RG. New horizons: Reablement - supporting older people towards independence. Age Ageing. 2016 Sep;45(5):572-6. doi: 10.1093/ageing/afw094. Epub 2016 May 21. PMID 27209329
- [Background] Age UK (2012) Day care services for elderly "hit by cuts". Reported by BBC news on 12th December 2012. bbc.co.uk/news/uk-20855819 Accessed on 28/06/2017.